CLINICAL TRIAL: NCT02697175
Title: Does Live Video Colposcopy Reduces Anxiety in Women With Cervical Dysplasia? A Randomised Trial.
Brief Title: Video Colposcopy in Women With Dysplasia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zydolab - Institute of Cytology and Immune Cytochemistry (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: COLPO-2
Record Dates: First submitted 2016-02-28; First posted 2016-03-03 (Estimated); Last update posted 2017-03-27 (Actual); Status verified 2017-03

CONDITIONS: Uterine Cervical Dysplasia
Keywords: live video-colposcopy; cervical dysplasia; anxiety; randomized controlled trial; colposcopy
MeSH Terms: conditions — Uterine Cervical Dysplasia; Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Live Video-Colposcopy (Experimental): Women are able to observe their colposcopic examination in real-time watching a flat screen in front of them
  Interventions: Device: Live Video-Colposcopy
- No Live Video-Colposcopy (Active Comparator): Women are not able to observe their colposcopic examination in real-time
  Interventions: Other: No Live Video-Colposcopy

INTERVENTIONS:
Device: Live Video-Colposcopy — The colposcopy will be shown in real time on a flat screen
  Arms: Live Video-Colposcopy
Other: No Live Video-Colposcopy — The TV will be shut off during colposcopy
  Arms: No Live Video-Colposcopy

SUMMARY:
To assess the effect of live video-colposcopy on women´s anxiety.

ELIGIBILITY:
Inclusion Criteria:

* women referred for colposcopy due to cervical abnormalities
* We included women if they attended colposcopy for the first time

Exclusion Criteria:

* pregnant women
* presence of a language barrier
* known anxiety disorder or depression
* history of conization or other treatments
* known oncological disorder
* inadequate colposcopy

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 275 (Actual)
Dates: Start 2016-08; Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Anxiety score after colposcopy | 10 minutes
  Each women completes the state anxiety questionnaire (state-trait anxiety inventory [STAI]) 10 minutes after colposcopy.

SECONDARY OUTCOMES:
Change in anxiety scores | 10 minutes
  Each women completes the state anxiety questionnaire (state-trait anxiety inventory [STAI]) before and 10 minutes after colposcopy. The difference in scores before and after colposcopy will be measured.
Pain during examination | 10 minutes
  women scores their pain level using a horizontal 100-mm visual analogue scale (VAS) ranging from 0 (,no pain') to 10 (,worst imaginable pain').
Pain after examination | 10 minutes
  women scores their pain level using a horizontal 100-mm visual analogue scale (VAS) ranging from 0 (,no pain') to 10 (,worst imaginable pain').
general unpleasantness during examination | 10 minutes
  women scores their feeeling during colposcopy using a horizontal 100-mm visual analogue scale (VAS) ranging from 0 ("not at all unpleasant") to 10 ("extremely unpleasant").
Anxiety during examination | 10 minutes
  women scores their anxiety during colposcopy using a horizontal 100-mm visual analogue scale (VAS) ranging from 0 ("no anxiety at all") to 10 ("worst imaginable anxiety")
Satisfaction concerning the medical consultation | 10 minutes
  women scores their satisfaction using a horizontal 100-mm visual analogue scale (VAS) ranging from 0 ("maximally unsatisfied") to 10 ("maximally satisfied").
Overall Satisfaction | 10 minutes
  women scores their satisfaction using a horizontal 100-mm visual analogue scale (VAS) ranging from 0 ("maximally unsatisfied") to 10 ("maximally satisfied").

CONTACTS AND LOCATIONS:
Overall Officials: Ziad Hilal, M.D., Principal Investigator — Zydolab - Institute of Cytology and Immune Cytochemistry
Locations (2):
- Germany (2):
  - Zydolab - Institute of Cytology and Immune Cytochemistry, Dortmund, North Rhine-Westphalia
  - Department of Obstetrics and Gynecology of the Ruhr University Bochum, Herne, North Rhine-Westphalia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hilal Z, Alici F, Tempfer CB, Seebacher V, Rezniczek GA. Video Colposcopy for Reducing Patient Anxiety During Colposcopy: A Randomized Controlled Trial. Obstet Gynecol. 2017 Aug;130(2):411-419. doi: 10.1097/AOG.0000000000002127. PMID 28697117